CLINICAL TRIAL: NCT04484636
Title: PLATON - Platform for Analyzing Targetable Tumor Mutations (Pilot-study) A Multicenter, Prospective, Cohort Study To Assess The Genomic Profiles And Associated Therapy Decision In Gastrointestinal Cancer
Brief Title: PLATON - Platform for Analyzing Targetable Tumor Mutations (Pilot-study)
Acronym: PLATON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PLATON pilot-study; AIO-HEP/STO-0219/ass (Other: AIO Arbeitsgemeinschaft Internistische Onkologie)
Record Dates: First submitted 2020-07-10; First posted 2020-07-23 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Cancer; Cholangiocarcinoma; Gallbladder Cancer; Pancreatic Cancer; Oesophageal Cancer; Stomach Cancer
Keywords: Gastric cancer; Individualized cancer therapy; Targetable mutations; Foundation Medicine assays; Hepatocellular Cancer; Cholangiocarcinoma; Gallbladder Cancer; Pancreatic Cancer; Oesophageal Cancer; Stomach Cancer; Platform-Design; Biobanking
MeSH Terms: conditions — Liver Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Experimental Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Hepatocellular Cancer (Other): molecular profiling - hepatocellular cancer (HCC)
  Interventions: Diagnostic Test: FoundationOne®CDx and FoundationOne®Liquid
- Cholangiocarcinoma (Other): molecular profiling - intra- and extrahepatic cholangiocellular carcinoma (CCA)
  Interventions: Diagnostic Test: FoundationOne®CDx and FoundationOne®Liquid
- Gallbladder Cancer (Other): molecular profiling - gallbladder carcinoma (GBCA)
  Interventions: Diagnostic Test: FoundationOne®CDx and FoundationOne®Liquid
- Pancreatic Cancer (Other): molecular profiling - pancreatic cancer (PanCa)
  Interventions: Diagnostic Test: FoundationOne®CDx and FoundationOne®Liquid
- Oesophageal Cancer + Stomach Cancer (Other): molecular profiling - esophagogastric cancer (EC/GC)
  Interventions: Diagnostic Test: FoundationOne®CDx and FoundationOne®Liquid

INTERVENTIONS:
Diagnostic Test: FoundationOne®CDx and FoundationOne®Liquid — FoundationOne CDx is a FDA-approved broad companion diagnostic (CDx) that is clinically and analytically validated for solid tumors. The test is designed to provide physicians with clinically actionable information - both to consider appropriate therapies for patients and understand results with evidence of resistance - based on the individual genomic profile of each patient's cancer. Every test result includes microsatellite instability (MSI) and tumor mutational burden (TMB) to help inform immunotherapy decisions. FoundationOne®Liquid is a liquid biopsy test for solid tumors that analyzes circulating tumor DNA (ctDNA) in blood.

SUMMARY:
PLATON (Platform for Analyzing Targetable Mutations) is a prospective, multicentre, observational cohort study with biobanking. In a first approach PLATON's pilot-study assesses genomic profiling in gastrointestinal cancer therapy and the frequencies of targetable mutations including Tumor Mutational Burden (TMB) and Microsatellite Instability Status (MSI), performing Next-generation deep sequencing (NGS) using the Foundation Medicine assays on tumor specimen and EDTA-whole blood samples. The Study Protocol does not define any further medical intervention or evaluate the efficacy or safety of the treatment decision made by the investigator. Another important objective of PLATON's pilot project is to evaluate whether and how many patients are treated based on their genomic profiles.

DETAILED DESCRIPTION:
PLATON (Platform for Analyzing Targetable Mutations) is designed to improve personalized therapy for patients in different cancer entities, such as in hepatocellular cancer (HCC), intra- and extrahepatic cholangiocellular carcinoma (CCA), gallbladder carcinoma (GBCA), pancreatic cancer (PanCa) and esophagogastric cancer (EC/GC), and elevate the treatment guidance within its framework. The key to understand the mechanisms in initiation, progression and response to treatment of cancer is the data integration of genetic mutational signatures with medical and physiological data of diseased cohorts.

PLATON is a prospective, multicentre, observational cohort study with biobanking and does not define any medical intervention or evaluate the efficacy or safety of the treatment decision made by the investigator.In a first approach PLATON's pilot-study assess genomic profiling in gastrointestinal cancer therapy and the frequencies of targetable mutations including Tumor Mutational Burden (TMB) and Microsatellite Instability Status (MSI), performing Next-generation deep sequencing (NGS) using the Foundation Medicine assays on tumor specimen and EDTA-whole blood samples. Another important objective of PLATON's pilot project is to evaluate whether and how many patients are treated based on their genomic profiles.

The pilot-study starts with the national-wide enrolment of 200 participants of both sexes and ages over 18 at 40 german study sites. The long-term vision is to enable cancer patients to receive the best available, scientifically founded, biomarker-based care, tailored to his or her individual needs

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of hepatocellular carcinoma or intra-/extrahepatic cholangiocarcinoma or gallbladder carcinoma or pancreatic ductal adenocarcinoma or esophagogastric adenocarcinoma in the advanced setting and no local curative therapy available.
* Standard first line therapy is planned, or patient is currently receiving first line therapy (started within the last 2 months before enrolment)
* ECOG 0-2
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Not able to understand all implications of study participation
* No written informed consent
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Distribution of mutations in patients with HCC, intra- and extrahepatic CCA, GBCA, PDAC and gastric cancer | up to 4 weeks after biospecimen provision
  Relative frequency of targetable mutations (incl. TMB and MSI status) computed as the number of patients who harbors at least one mutation divided by the number of total patients in the pooled patient population.

SECONDARY OUTCOMES:
Heterogeneity of targetable alterations in paraffin embedded specimen vs. cfDNA | up to 4 weeks after biospecimen provision
  Number of differences (heterogeneity) in targetable alterations in paraffin specimen vs. cfDNA
Relative frequency of targetable mutations (incl. TMB and MSI status) per disease group | up to 4 weeks after biospecimen provision
  Relative frequency of targetable mutations (incl. TMB and MSI status) per disease group
Number of patients receiving therapies in accordance to their genomic profiles | up to 4 weeks after biospecimen provision
  Number of patients receiving therapies in accordance to their genomic profiles

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Arndt Vogel, Prof., Principal Investigator — Hannover Medical School
Locations (46):
- Germany (46):
  - KHNW Frankfurt, Frankfurt am Main, Hesse
  - Hannover Medical School, Hanover, Lower Saxony
  - Onkologische Schwerpunktpraxis Speyer, Speyer, Rhineland-Palatinate
  - Elblandklinikum Riesa, Ried, Saxony
  - Friedrich-Ebert-Krankenhaus Neumünster, Neumünster, Schleswig-Holstein
  - MVZ Oskar-Helene-Heim Berlin, Berlin, State of Berlin
  - Sana Kliniken Leipziger Land, Borna, Thuringia
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Klinikum Bayreuth, Bayreuth
  - Vivantes Klinikum Spandau, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Augusta-Kranken-Anstalt Bochum, Bochum
  - Bochum Uni, Bochum
  - Klinikum Chemnitz, Chemnitz
  - Klinikum Darmstadt, Darmstadt
  - GEFOS - Gesellschaft für onkologische Studien Dortmund, Dortmund
  - Onkozentrum Dresden, Dresden
  - Klinikum Frankfurt Höchst, Frankfurt
  - Klinikum Fulda, Fulda
  - MVZ Onkologische Kooperation Harz, Goslar
  - Universitätsklinikum Halle (Saale), Halle
  - Hamburg Onkologisch-Hämatologische Schwerpunktpraxis, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - St. Anna Hospital Herne, Herne
  - Ortenau Klinikum Lahr-Ettenheim, Lahr
  - ÜBAG - MVZ Dr. Vehling-Kaiser GmbH, Landshut
  - Langen, Gemeinschaftspraxis für Hämatologie und Onkologie, Langen
  - Studienzentrum UnterEms, Leer
  - Klinikum Lippe, Lemgo
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsklinikum Giessen und Marburg GmbH, Marburg
  - Klinik München-Bogenhausen, München
  - Münster, Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Niels-Stensen-Kliniken Osnabrück, Osnabrück
  - Medius Klinik Osterfildern-Ruit, Ostfildern
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Klinikum Rheine, Mathias-Spital Rheine, Rheine
  - RoMed Klinikum Rosenheim, Rosenheim
  - Klinikum Südstadt Rostock, Rostock
  - CaritasKlinikum Saarbrücken, Saarbrücken
  - Onkologie Bodensee, Singen
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH, Wiesbaden
  - Marien Hospital Witten, Witten
  - Klinikum Wolfsburg, Wolfsburg
  - Onkologisches Zentrum Wolfsburg-Helmstedt MVZ GmbH, Wolfsburg

IPD SHARING:
Plan to Share IPD: No
Depending on particpant informed concent individual-participant data (IPD) will only be shared in research-cooperations according the terms of PLATON's Use and Access Regulation. Scientific projects have to be approved by PLATON'S Scientific Steering Committee.

REFERENCES:
- See also: The PLATON Network — https://platon-network.de/